CLINICAL TRIAL: NCT04889950
Title: A Randomized, Masked (Evaluator), Controlled, Prospective Pilot Study of the Effectiveness and Safety of the Tixel Versus Lipiflow in the Treatment of Meibomian Gland Dysfunction.
Brief Title: Evaluate the Safety and Effectiveness of The Tixel Fractional System in the Treatment of Meibomian Gland Disfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Novoxel Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLN 0798
Record Dates: First submitted 2021-05-03; First posted 2021-05-17 (Actual); Results first posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Dry Eye Syndromes; Dry Eye; Meibomian Gland Dysfunction
MeSH Terms: conditions — Dry Eye Syndromes; Meibomian Gland Dysfunction

STUDY DESIGN:
Intervention Model Description: A Randomized, Masked (Evaluator), Controlled, Prospective Pilot Study
Who Masked: Outcomes Assessor
Masking Description: Blinded Evaluator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tixel Group (Experimental): Tixel C Group: Screening and baseline visits, Treatment- 3 treatment sessions, followed by 2 Follow up sessions, 1and 3 months after last treatment visit. Subject will be questioned about Discomfort and Pain Questionnaires (self-assessed) and OSDI questionnaire.
  Interventions: Device: Tixel C
- LipiFlow (Active Comparator): LipiFlow: Screening and baseline visits, Treatment- 1 single treatment session, followed by 2 Follow up sessions, 1and 3 months after the last treatment visit. Subject will be questioned about Discomfort and Pain Questionnaires (self-assessed) and OSDI questionnaire.
  Interventions: Device: LipiFlow

INTERVENTIONS:
Device: Tixel C — Tixel C )Novoxel®, Israel) is a thermomechanical system developed for fractional treatment. The system is designed for the treatment of soft tissue by direct conduction of heat, enabling tissue coagulation combined with micro ablation with low thermal damage to the surrounding tissue.
  Arms: Tixel Group
Device: LipiFlow — LipiFlow
  Arms: LipiFlow

SUMMARY:
A Randomized, Masked (Evaluator), Controlled, Prospective Pilot Study of the Effectiveness and Safety of the Tixel®, Versus LipiFlow® in the Treatment of Meibomian Gland Dysfunction. Up to 30 patients (60 eyes) to be randomized in up to 2 clinical sites in Israel and/or Europe. study subject will receive three (3) treatments with Tixel in a monthly interval, and a single treatment for the control group. Follow-up will occur 1 month and 3 months following the last treatment.

DETAILED DESCRIPTION:
Up to 30 patients (60 eyes), 15 Per Device at up to 2 study sites in Israel and/or Europe will be recruited to evaluate the safety and effectiveness of the Tixel device in adults with Meibomian Gland Dysfunction (MGD). study subject will receive three (3) treatments with Tixel in a monthly interval, and single treatment for the control group. Follow-up will occur 1 month and 3 months following the last treatment.

Tixel group study visits will be as follow:

Screening: (Must be done up to 7 days prior to initial treatment (Day 0), but can be also done on the same day as baseline testing and initial treatment) Randomization: (Performed after determining that patient is eligible for the study) Treatments - three treatments will be conducted to the study device group. Follow-Up Visits: 4-Weeks (+/-7days) and 12-Weeks (+/-14 days) after last treatment.

Control group visit will be as follow:

Screening: (Must be done up to 7 days prior to initial treatment (Day 0), but can be also done on the same day as baseline testing and initial treatment) Randomization: (Performed after determining that patient is eligible for the study) Treatment- single Follow-Up Visits: 4-Weeks (+/-7days) and 12-Weeks (+/-14 days) after last treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older of any gender or race.
* Provision of written informed consent prior to study participation.
* Willingness and ability to return for all study visits.
* A positive history of self-reported dry eye symptoms for three months prior to the study using the Ocular Surface Disease Index (OSDI) questionnaire, and a score of ≥ 23 at the baseline visit.
* Evidence of meibomian gland (MG) obstruction, based on a total Meibomian Gland Score (MGS) of ≤12 in the lower eyelids for each eye. The rater of MGS must not be involved in the study procedure.
* Tear break-up time (TBUT) <10 seconds. The rater of TBUT must not be involved in the study procedure.
* Agreement/ability to abstain from dry eye/MGD medications for the time between the treatment visit/s and the final study visit. Ocular lubricants are allowed if no changes are made during the study.
* Fitzpatrick skin type I-VI

Exclusion Criteria:

* History of ocular surgery including intraocular, oculo-plastic, corneal or refractive surgery within 1 year.
* Patients with giant papillary conjunctivitis.
* Patients with punctal plugs or who have had punctal cautery.
* Ocular injury or trauma, chemical burns, or limbal stem cell deficiency within 3 months of the baseline examination.
* Active ocular herpes zoster or simplex of eye or eyelid or a history of these within the last 3 months.
* Patients who are aphakic.
* Cicatricial lid margin disease identified via slit lamp examination, including pemphigoid, symblepharon, etc.
* Active ocular infection (e.g., viral, bacterial, mycobacterial, protozoan, or fungal infection of the cornea, conjunctiva, lacrimal gland, lacrimal sac, or eyelids including a hordeolum or stye).
* Active ocular inflammation or history of chronic, recurrent ocular inflammation within prior 3 months (e.g. retinitis, macular inflammation, choroiditis, uveitis, iritis, scleritis, episcleritis, keratitis).
* Ocular surface abnormality that may compromise corneal integrity (e.g., prior chemical burn, recurrent corneal erosion, corneal epithelial defect, Grade 3 corneal fluorescein staining, or map dot fingerprint dystrophy).
* Lid surface abnormalities (e.g., entropion, ectropion, tumor, edema, blepharospasm, lagophthalmos, severe trichiasis, severe ptosis) that may affect lid function in either eye.
* Anterior blepharitis (staphylococcal, demodex, or seborrheic grade 3 or 4).
* Systemic disease conditions that cause dry eye (e.g., Stevens- Johnson syndrome, vitamin A deficiency, rheumatoid arthritis, Wegener's granulomatosis, sarcoidosis, leukemia, Riley-Day syndrome, systemic lupus erythematosus, Sjogren's syndrome).
* Unwillingness to abstain from systemic medications known to cause dryness for the study duration.
* Women in child bearing age who are pregnant, nursing, or not utilizing adequate birth control measures.
* Individuals who have changed the dosing of either systemic or non-dry eye/MGD ophthalmic medication within the past 30 days prior to screening.
* Individuals who are unable or unwilling to remain on a stable dosing regimen for the duration of the study.
* Individuals using isotretinoin (Accutane) within 1 year, cyclosporine-A (Restasis) or lifitegrast ophthalmic solution (Xiidra) within 3 months, or any other dry eye or MGD medications (antibiotics, non-steroidal anti-inflammatory drugs, corticosteroids) for at least 2weeks; and to maintain abstinence throughout the duration of the study (ocular lubricants are allowed if no changes are made during the study).
* Individuals wearing contact lenses at any time during the prior three months and at any point during the study.
* Current skin cancer, malignant sites and/or advanced premalignant lesions or moles in the treatment area.
* An impaired immune system condition or use of immunosuppressive medication.
* Collagen disorders, keloid formation and/or abnormal wound healing.
* Previous invasive/ablative procedures in the areas to be treated within 3 months prior to initial treatment or plans for such treatment during the course treatment, or before complete healing of such treatments has occurred.
* Any patient who takes or has taken any oral or topical medications, herbal treatment, food supplements, or vitamins which may cause fragile skin or impaired skin healing during the last 3 months.
* Any patient who has a history of bleeding coagulopathies.
* Any patient who has tattoos or permanent makeup in the treated area.
* Any patient who has burned, blistered, irritated or sensitive skin in any of the areas to be treated.
* Individuals using another ophthalmic investigational device or agent within 30 days of study participation.
* Individuals that were treated in either eye with LipiFlow in the last 24 months, or Tixel at any point in the past.
* Treatment in either eye with IPL in the last year.
* Expression of the meibomian glands within 6 months prior to screening.
* Use of at home warm compresses or lid hygiene products while participating in study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-10-26 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2023-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ehud Reich, MD, Principal Investigator — Shaare Zedek Medical Center
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: eyes
Groups:
- Tixel Group: Tixel C Group: Screening and baseline visits, Treatment- 3 treatment sessions, followed by 2 Follow up sessions, 1and 3 months after last treatment visit. Subject will be questioned about Discomfort and Pain Questionnaires (self-assessed) and OSDI questionnaire.
  Tixel C: Tixel C (Novoxel®, Israel) is a thermomechanical system developed for fractional treatment. The system is designed for the treatment of soft tissue by direct conduction of heat, enabling tissue coagulation combined with micro ablation with low thermal damage to the surrounding tissue.
Period: Overall Study
Arm/Group | Tixel Group | LipiFlow
Started | 11; 22 eyes (subjects) | 10; 20 eyes (subjects)
Completed | 9; 18 eyes (subjects) | 10; 20 eyes (subjects)
Not Completed | 2; 4 eyes | 0; 0 eyes

BASELINE CHARACTERISTICS:
Population: study subjects comparing the Tixel device to LipiFlow System
Groups:
- Total: Total of all reporting groups
Arm/Group | Tixel Group | LipiFlow | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 8 | 15
  >=65 years | 4 | 2 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (18.9) | 59.4 (7.7) | 58.4 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 2 | 3 | 5
Race/Ethnicity, Customized [Number; unit: participants]
  caucasian | 11 | 8 | 19
  white | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Israel | 11 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: Score and Change From Baseline in Tear Break Up Times (TBUT), as Assessed by a Masked Rater
Description: Change from baseline to the 4-weeks follow-up exam in Tear Break Up Times (TBUT), as assessed by a masked rater.
  TBUT - Tear Break-Up Time, is a clinical test used to evaluate the stability of the tear film on the surface of the eye. It measures the time it takes for dry spots to appear on the cornea after a blink. A shorter TBUT indicates a more unstable tear film, which can be a sign of dry eye disease or other ocular surface disorders.
  Tear Break-Up Time (TBUT) is typically scored by the time (in seconds). The general interpretation of TBUT scores is as follows:
  Normal TBUT: More than 10 seconds Borderline TBUT: 5 to 10 seconds Abnormal/Low TBUT: Less than 5 seconds
Time Frame: Tixel arm: Baseline and 4 weeks after last treatment (8 weeks post baseline). LipiFlow arm: Baseline and 4 weeks after treatment (4 weeks post baseline).
Population: 10 Tixel subjects and 10 LipiFlow subjects completed the Baseline and 4-week FU TBUT examination.
Measure: Mean (95% Confidence Interval); unit: seconds
Units Other Than Participants: Eyes
Arm/Group | Tixel Group | LipiFlow
Number analyzed (Participants) | 10 | 10
Number analyzed (Eyes) | 20 | 20
seconds
  4 weeks change from baseline | 4.0 [2.3 to 5.6] | 1.9 [0.8 to 3.0]
  Baseline score | 3.4 [3.1 to 3.7] | 4.7 [3.9 to 5.4]
  4 weeks FU score | 7.4 [5.8 to 9.1] | 6.6 [5.3 to 7.8]

2. Primary Outcome: Comparison of the Incidence of Device-related Adverse Events for the Two-treatment Arms.
Description: Comparison of the incidence of device-related adverse events (e.g., increase in the lid margin such as development of floppy eyelids, entropion or ectropion; and lash integrity) for the two-treatment arms.
Time Frame: Tixel arm: Baseline to 12 weeks after last treatment (16 weeks post baseline). LipiFlow arm: Baseline to 12 weeks after treatment (12 weeks post baseline).
Population: Ae's observed in Tixel group compared to Lipiflow group
Measure: Number; unit: number of events
Arm/Group | Tixel Group | LipiFlow
Number analyzed (Participants) | 11 | 10
number of events | 0 | 0

3. Secondary Outcome: Score on a Scale and Change From Baseline in Patient Symptoms Using Ocular Surface Disease Index (OSDI).
Description: Change from baseline in patient symptoms using Ocular Surface Disease Index (OSDI) at 4-weeks and 12-weeks follow-up exam.
  The Ocular Surface Disease Index (OSDI) is a questionnaire designed to assess the severity of dry eye disease.
  OSDI Questionnaire
  The questionnaire consists of 12 questions divided into three subscales:
  Ocular Symptoms Visual Functioning Environmental Triggers
  Scoring System
  The scoring for the OSDI is based on a scale from 0 to 100, where higher scores indicate more severe symptoms. Each question is scored as follows:
  0: None of the time
  1. Some of the time
  2. Half of the time
  3. Most of the time
  4. All of the time
  Interpretation of OSDI Scores
  The OSDI scores are generally interpreted as follows:
  0-12: Normal or no dry eye 13-22: Mild dry eye 23-32: Moderate dry eye 33-100: Severe dry eye
Time Frame: as for outcome 2
Population: Tixel subects and lipiflow subjects completed baseline, 4 weeks OSDI and 12 weeks OSDI.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | Tixel Group | LipiFlow
Number analyzed (Participants) | 10 | 10
Number analyzed (Eyes) | 20 | 20
score on a scale
  OSDI at Baseline | 42.7 [30.4 to 55.0] | 47.6 [33.8 to 61.4]
  OSDI at 4 weeks | 22.0 [10.0 to 34.0] | 38.2 [19.2 to 57.3]
  OSDI at 12 weeks: number analyzed (Participants) | 9 | 10
  OSDI at 12 weeks: number analyzed (Eyes) | 18 | 20
  OSDI at 12 weeks | 27.0 [10.7 to 43.3] | 32.4 [17.1 to 47.8]
  change from baseline to 4 weeks | -20.7 [-25.5 to -15.9] | -9.4 [-22.7 to 3.9]
  change from baseline at 12 weeks FU: number analyzed (Participants) | 9 | 10
  change from baseline at 12 weeks FU: number analyzed (Eyes) | 18 | 20
  change from baseline at 12 weeks FU | -15.4 [-27.4 to -3.4] | -15.2 [-28.4 to -1.9]

4. Secondary Outcome: Score on a Scale and Change From Baseline in Meibomian Gland Score (MGS), as Assessed by a Masked Rater.
Description: score on a scale at baseline, 4-weeks and 12-weeks follow-up exam in Meibomian Gland (MGS), as assessed by a masked rater.
  The Meibomian Gland Score (MGS) is a clinical tool used to evaluate the function of the meibomian glands.
  Scoring Criteria
  Each gland is assessed and scored based on the quality of the expressed secretion:
  0: No secretion
  1. Inspissated
  2. Cloudy
  3. Clear liquid
  Interpretation of MGS Minimal MGS score = 0 in each eye (15 glands evaluated in each eye) Maximal MGS score = 45 in each eye (15 glands evaluated in each eye) Low MGS: (below 12) Indicates poor function or obstruction of the meibomian glands, suggesting MGD.
Time Frame: as for outcome 2
Population: subject in the tixel group and subject in the lipiflow group comparisoon at baseline, 4 weeks and 12 weeks visits.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | Tixel Group | LipiFlow
Number analyzed (Participants) | 10 | 10
Number analyzed (Eyes) | 20 | 20
score on a scale
  MGS at baseline | 2.5 [1.0 to 4.0] | 4.5 [2.9 to 6.1]
  MGS at 4 weeks | 13.7 [7.6 to 19.7] | 5.6 [3.0 to 8.2]
  MGS at 12 weeks: number analyzed (Participants) | 9 | 10
  MGS at 12 weeks: number analyzed (Eyes) | 18 | 20
  MGS at 12 weeks | 9.8 [4.5 to 15.1] | 13.9 [9.0 to 18.7]
  4 weeks MGS Change from Baseline | 11.2 [5.3 to 17.0] | 1.1 [-1.6 to 3.8]
  12 weeks MGS Change from Baseline: number analyzed (Participants) | 9 | 10
  12 weeks MGS Change from Baseline: number analyzed (Eyes) | 18 | 20
  12 weeks MGS Change from Baseline | 7.1 [1.4 to 12.8] | 9.4 [4.8 to 13.9]

5. Secondary Outcome: Overall Changes From Baseline in Tear Break Up Times (TBUT), as Assessed by a Masked Rater.
Description: Changes from baseline to the 12-weeks follow-up exam in Tear Break Up Times (TBUT), as assessed by a masked rater.
  BUT - Tear Break-Up Time, is a clinical test used to evaluate the stability of the tear film on the surface of the eye. It measures the time it takes for dry spots to appear on the cornea after a blink. A shorter TBUT indicates a more unstable tear film, which can be a sign of dry eye disease or other ocular surface disorders.
  Tear Break-Up Time (TBUT) is typically scored by the time (in seconds). The general interpretation of TBUT scores is as follows:
  Normal TBUT: More than 10 seconds Borderline TBUT: 5 to 10 seconds Abnormal/Low TBUT: Less than 5 seconds
Time Frame: Tixel arm: Baseline and 12 weeks after last treatment (16 weeks post baseline). LipiFlow arm: Baseline and 12 weeks after treatment (12 weeks post baseline).
Population: 9 Tixel subjects and 10 LipiFlow subjects completed the 12-week FU TBUT examination.
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: Eyes
Arm/Group | Tixel Group | LipiFlow
Number analyzed (Participants) | 9 | 10
Number analyzed (Eyes) | 18 | 20
seconds | 4.2 (2.9) | 1.6 (2.2)

6. Secondary Outcome: Score on a Scale During Treatment Discomfort and Pain Questionnaires (Each Self-assessed by VAS)
Description: Discomfort and Pain from the treatment (Tixel or LipiFlow) using the questionnaires assessed by the subject. These are visual analogue scale (VAS) questionnaires using a scale from 0-10 to assess eye discomfort and pain. Both questionnaires are to be self-assessed by the patient immediately following treatment.
  Interpetation for the assessment:
  score 0- no discomfort / pain score 5 - moderate discomfort / pain score 10 - worst possible discomfort / pain
Time Frame: Tixel arm: 4 weeks (treatment 1- day 0, treatment 2- 2 weeks, treatment 3- 4 weeks). LipiFlow arm: On treatment day - day 0 (only one treatment for this arm)
Population: Post-Treatment Pain Questionnaire scores, by tixel and lipiflow groups
Measure: Mean (95% Confidence Interval); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | Tixel Group | LipiFlow
Number analyzed (Participants) | 11 | 10
Number analyzed (Eyes) | 22 | 20
score on a scale
  post Treatment 1 pain score | 3.9 [2.6 to 5.3] | 0.5 [0.1 to 1.0]
  post Treatment 2 pain score: number analyzed (Participants) | 10 | 0
  post Treatment 2 pain score: number analyzed (Eyes) | 20 | 0
  post Treatment 2 pain score | 3.6 [2.6 to 4.6] |
  post Treatment 3 pain score: number analyzed (Participants) | 10 | 0
  post Treatment 3 pain score: number analyzed (Eyes) | 20 | 0
  post Treatment 3 pain score | 2.8 [2.2 to 3.4] |
  post Treatment 1 discomfort score | 3.7 [2.5 to 4.9] | 0.9 [0.2 to 1.5]
  post Treatment 2 discomfort score: number analyzed (Participants) | 10 | 0
  post Treatment 2 discomfort score: number analyzed (Eyes) | 20 | 0
  post Treatment 2 discomfort score | 3.6 [2.5 to 4.7] |
  post Treatment 3 discomfort score: number analyzed (Participants) | 10 | 0
  post Treatment 3 discomfort score: number analyzed (Eyes) | 20 | 0
  post Treatment 3 discomfort score | 3.6 [2.7 to 4.4] |

7. Secondary Outcome: Corneal Fluorescein Staining Slit Lamp Evaluation Scores and Change From Baseline
Description: Changes from baseline following treatment for the test and control devices for the following assessments:
  Ocular Surface Staining (to evaluate the integrity of the corneal epithelium by identifying areas of damage or staining)
  Grading scale:
  0 = Normal - No staining
  1. = Mild - Superficial stippling micropunctate staining
  2. = Moderate - Macropunctate staining with some coalescent areas
  3. = Severe - Numerous coalescent macropunctate areas and/or patches
  5 regions (superior, temporal, central, nasal, and inferior) are graded for each eye. total score range from 0 -15.
Time Frame: as for outcome 2
Population: Corneal Fluorescein Staining Slit Lamp evaluation score (Safety population)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | Tixel Group | LipiFlow
Number analyzed (Participants) | 11 | 10
Number analyzed (Eyes) | 22 | 20
score on a scale
  Baseline score | 6.6 [4.9 to 8.4] | 3.6 [1.8 to 5.3]
  Treatment 1 score | 6.6 [4.9 to 8.3] | 3.6 [2.1 to 5.1]
  treatment 2 score: number analyzed (Participants) | 10 | 0
  treatment 2 score: number analyzed (Eyes) | 20 | 0
  treatment 2 score | 2.0 [1.1 to 2.8] |
  treatment 3 score: number analyzed (Participants) | 10 | 0
  treatment 3 score: number analyzed (Eyes) | 20 | 0
  treatment 3 score | 1.2 [0.4 to 1.9] |
  4 weeks FU score: number analyzed (Participants) | 10 | 10
  4 weeks FU score: number analyzed (Eyes) | 20 | 20
  4 weeks FU score | 2.1 [0.7 to 3.4] | 2.4 [1.5 to 3.3]
  12 weeks FU score: number analyzed (Participants) | 9 | 10
  12 weeks FU score: number analyzed (Eyes) | 18 | 20
  12 weeks FU score | 2.0 [1.1 to 2.9] | 1.8 [0.5 to 3.1]
  Treatment 1 change from baseline | -0.0 [-1.0 to 0.9] | 0.1 [-1.5 to 1.6]
  Treatment 2 change from baseline: number analyzed (Participants) | 10 | 0
  Treatment 2 change from baseline: number analyzed (Eyes) | 20 | 0
  Treatment 2 change from baseline | -4.3 [-6.0 to -2.5] |
  Treatment 3 change from baseline: number analyzed (Participants) | 10 | 0
  Treatment 3 change from baseline: number analyzed (Eyes) | 20 | 0
  Treatment 3 change from baseline | -5.1 [-6.4 to -3.7] |
  4 weeks FU change from baseline: number analyzed (Participants) | 10 | 10
  4 weeks FU change from baseline: number analyzed (Eyes) | 20 | 20
  4 weeks FU change from baseline | -4.2 [-5.9 to -2.4] | -1.2 [-3.0 to 0.7]
  12 weeks FU change from baseline: number analyzed (Participants) | 9 | 10
  12 weeks FU change from baseline: number analyzed (Eyes) | 18 | 20
  12 weeks FU change from baseline | -3.8 [-5.6 to -1.9] | -1.8 [-2.7 to -0.8]

8. Secondary Outcome: The Mean Changes From Baseline in IOP for All Eyes on the Tixel and Lipiflow Arms
Description: the IOP values changes from baseline, respectively, for all visits, per treatment arm.
Time Frame: as for outcome 2
Population: IOP values in mmHg and the changes from baseline to 12 weeks FU
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: Eyes
Arm/Group | Tixel Group | LipiFlow
Number analyzed (Participants) | 11 | 10
Number analyzed (Eyes) | 22 | 20
mmHg
  Treatment 1 | -0.3 (3.0) | -3.3 (2.2)
  Treament 2: number analyzed (Participants) | 10 | 0
  Treament 2: number analyzed (Eyes) | 20 | 0
  Treament 2 | -1.5 (2.5) |
  Treatment 3: number analyzed (Participants) | 10 | 0
  Treatment 3: number analyzed (Eyes) | 20 | 0
  Treatment 3 | -1.5 (2.0) |
  4 weeks FU: number analyzed (Participants) | 10 | 10
  4 weeks FU: number analyzed (Eyes) | 20 | 20
  4 weeks FU | 0.2 (2.8) | -0.1 (2.0)
  12 weeks FU: number analyzed (Participants) | 9 | 10
  12 weeks FU: number analyzed (Eyes) | 18 | 20
  12 weeks FU | 0.4 (2.3) | 1.5 (2.1)

9. Secondary Outcome: Lissamine Green Staining Scores and the Changes From Baseline
Description: Changes from baseline following treatment for the test and control devices for the following assessments:
  Lissamine staining scores (to assess the health of the conjunctival and corneal epithelium, particularly in dry eye disease, by identifying areas of damaged or dead cells).
  Grading scale:
  0 = Normal - No staining
  1. = Mild - Superficial stippling micropunctate staining
  2. = Moderate - Macropunctate staining with some coalescent areas
  3. = Severe - Numerous coalescent macropunctate areas and/or patches
  6 regions (nasal, superior nasal, inferior nasal, temporal, superior temporal, inferior temporal) are graded for each eye. total score range for each eye is 0-18.
Time Frame: as for outcome 2
Population: subjects performed Lissamine staining scoresat baseline and during study visits
Measure: Mean (95% Confidence Interval); unit: score on a scale
Units Other Than Participants: Eyes
Arm/Group | Tixel Group | LipiFlow
Number analyzed (Participants) | 11 | 10
Number analyzed (Eyes) | 22 | 20
score on a scale
  Baseline | 6.1 [5.0 to 7.3] | 4.7 [3.4 to 6.0]
  Treatment 1 | 5.4 [4.0 to 6.8] | 3.1 [2.0 to 4.1]
  Treatment 2: number analyzed (Participants) | 10 | 0
  Treatment 2: number analyzed (Eyes) | 20 | 0
  Treatment 2 | 1.5 [0.7 to 2.2] |
  Treatment 3: number analyzed (Participants) | 10 | 0
  Treatment 3: number analyzed (Eyes) | 20 | 0
  Treatment 3 | 1.0 [0.2 to 1.8] |
  4 weeks FU: number analyzed (Participants) | 10 | 10
  4 weeks FU: number analyzed (Eyes) | 20 | 20
  4 weeks FU | 1.4 [0.4 to 2.3] | 3.3 [2.2 to 4.4]
  12 weeks FU: number analyzed (Participants) | 9 | 10
  12 weeks FU: number analyzed (Eyes) | 18 | 20
  12 weeks FU | 1.9 [0.7 to 3.0] | 1.5 [0.4 to 2.6]
  Treatment 1 change from baseline | -0.7 [-1.5 to 0.0] | -1.7 [-2.7 to -0.6]
  Treatment 2 change from baseline: number analyzed (Participants) | 10 | 0
  Treatment 2 change from baseline: number analyzed (Eyes) | 20 | 0
  Treatment 2 change from baseline | -4.9 [-6.2 to -3.6] |
  Treatment 3 change from baseline: number analyzed (Participants) | 10 | 0
  Treatment 3 change from baseline: number analyzed (Eyes) | 20 | 0
  Treatment 3 change from baseline | -5.4 [-6.7 to -4.0] |
  FU 4 weeks change from baseline: number analyzed (Participants) | 10 | 10
  FU 4 weeks change from baseline: number analyzed (Eyes) | 20 | 20
  FU 4 weeks change from baseline | -5.0 [-6.4 to -3.6] | -1.4 [-3.0 to 0.2]
  FU 12 weeks change from baseline: number analyzed (Participants) | 9 | 10
  FU 12 weeks change from baseline: number analyzed (Eyes) | 18 | 20
  FU 12 weeks change from baseline | -4.1 [-5.8 to -2.3] | -3.2 [-4.7 to -1.7]

ADVERSE EVENTS:
Time Frame: 15 months and 13 days
Description: A total of 12 device not related AEs were observed in 7 subjects (4 Tixel subjects (3.6%) and 3 (3%) LipiFlow subjects). One moderate AE ('Conjunctival deposit') was reported in one subject and resolved after medication administration and removal of conjunctival concretions. All other AEs were mild and resolved.
Arm/Group | Tixel Group | LipiFlow
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 4/11 | 3/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tixel Group (N=11) | LipiFlow (N=10)
Conjunctival deposit (Eye disorders) | 1 (2) | 0 (0) — Conjunctival deposit
Corneal opacity (Eye disorders) | 1 (1) | 0 (0) — Corneal opacity
COVID-19 (Infections and infestations) | 1 (1) | 2 (2) — COVID-19
Pulpitis dental (Infections and infestations) | 1 (1) | 0 (0) — Pulpitis dental
Conjunctival scar (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Conjunctival scar
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Intervertebral disc protrusion
Migraine (Nervous system disorders) | 1 (1) | 0 (0) — Migraine
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Rash papular
Chalazion (Eye disorders) | 1 (1) | 0 (0) — Chalazion

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-21): https://cdn.clinicaltrials.gov/large-docs/50/NCT04889950/Prot_SAP_000.pdf